CLINICAL TRIAL: NCT01653184
Title: The Effect of Oral Supplementation With Omega-3 Fatty Acids on Serum Omega-3 Levels in Patients With Age-related Macular Degeneration: A Randomized Controlled Trial.
Brief Title: Effect of Omega-3-fatty Acids on Blood Levels Omega-3 Fatty Acids in Patients With Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Physician Recommended Nutriceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Omega 20120660; Protocol #20120660 (Other: WIRB)
Record Dates: First submitted 2012-07-25; First posted 2012-07-30 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Macular Degeneration
Keywords: AMD; Vision loss; omega-3; supplement; age related macular degeneration
MeSH Terms: conditions — Macular Degeneration; Vision Disorders | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: AREDS 2 Vitamin formula 1g (Experimental): Patients will receive oral supplementation with the commercially available "AREDS2" vitamin formula (PreserVision AREDS 2 Eye Vitamin and Mineral Supplement. Bausch + Lomb Incorporated), consisting of vitamins C, E, zinc, lutein, zeaxanthin and 1g of omega-3 fatty acids in the ethyl ester formulation
  Interventions: Dietary Supplement: Omega-3 fatty acid
- Eye Omega Advantage 2g (Experimental): Patients will receive a similar vitamin combination in the second arm (Eye Omega Advantage® and Macular Vitamin Benefit. Physician Recommended Nutriceuticals) with 2g of omega-3 fatty acids in the triglyceride formulation (see attached document for supplement details)
  Interventions: Dietary Supplement: Omega-3 fatty acid

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — The purpose of our study is to evaluate the change in serum omega-3 index (blood level of omega-3 fatty acids) after 1 gram of omega-3 fatty acid supplementation versus 2 grams.

SUMMARY:
The effect of omega-3-fatty acids on blood levels omega-3 fatty acids in patients with age-related macular degeneration.

DETAILED DESCRIPTION:
There is observational data in the current literature suggesting that the intake of foods high in marine sources of omega-3 fatty acids, such as fish, may lower the risk of developing age-related macular degeneration (AMD). A large prospective study is underway to determine whether oral supplementation with 1 gram of omega-3 fatty acids is beneficial for subjects with dry AMD. The purpose of our study is to evaluate the change in serum omega-3 index (blood level of omega-3 fatty acids) after 1 gram of omega-3 fatty acid supplementation versus 2 grams.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Have AREDS category 3 or 4 disease.
* Category 3: Many medium sized drusen or one or more large drusen in one or both eyes
* Category 4: Geographic atrophy or choroidal neovascularization in one eye.

Exclusion Criteria:

* Women of child-bearing age with positive urine pregnancy tests or desire to conceive during the course of the study.
* Patients with a known fish allergy.
* Patients currently taking supplementation with omega-3 fatty acids and have an omega-3 index of greater than 4%.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in omega-3 index | Monthly for 6 months
  To determine the change in omega-3 index using an omega-3 index serum test, in patients with dry AMD given the commercially available AREDS2 formula supplementation (containing 1gram of omega-3 fatty acids in ethyl ester formulation) compared to patients given a similar vitamin combination with 2 grams of omega-3 fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Fineman, MD, Principal Investigator — Mid Atlantic Retina
Locations (4):
- United States (4):
  - Mid Atlantic Retina- Cherry Hill, Cherry Hill, New Jersey
  - Mid Atlantic Retina - Bethlehem, Bethlehem, Pennsylvania
  - Mid Atlantic Retina- Hungtindon Valley, Huntingdon Valley, Pennsylvania
  - Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No